CLINICAL TRIAL: NCT02323217
Title: I2PETHV - Quantification and Localisation of Imidazoline2 Binding Sites in Healthy Volunteers Using [11C]BU99008 a Positron Emission Tomography Study
Brief Title: I2PETHV - Imidazoline2 Binding Site in Healthy Volunteers
Acronym: I2PETHV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14HH2250; MR/L01307X/1 (Other Grant/Funding Number: MRC)
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers; Alzheimer Disease; Molecular Imaging
Keywords: Imidazoline Receptor 2; (4,5-dihydro-1H-imidazol-2-yl)-1-methyl-1H-indole; BU99008; Radionuclide Imaging; Molecular Imaging; Healthy Volunteers; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Idazoxan; Isocarboxazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Experimental)
  Interventions: Radiation: [11C]BU99008; Drug: Idazoxan; Drug: Isocarboxazid

INTERVENTIONS:
Radiation: [11C]BU99008 — Baseline Scan, Test-ReTest or Dosimetry
Drug: Idazoxan — Idazoxan block of [11C]BU99008
Drug: Isocarboxazid — Isocarboxazid block of [11C]BU99008

SUMMARY:
The imdazoline2 binding site (I2BS) is known to reside inside astrocytes. Changes in the numbers of I2BS in post mortem tissue has implicated them in a range of psychiatric conditions such as depression and addiction, along with neurodegenerative disorders such as Alzheimer's disease and Huntington's chorea. Preclinical studies have also demonstrated functional interactions with the opioid system, where I2BS ligands have been shown to affect tolerance to morphine and alleviate some of the morphine withdrawal syndrome in rats. Recently the I2BS and I2BS ligands have been shown to have some interesting analgesic effects in different models of pain and a novel I2BS ligand, CR4056, is currently undergoing Phase II clinical trials as a novel treatment for neuropathic pain and acute non- specific pain states.

The location of I2BS on astrocytic glial cells and the possibility that they may in some way regulate glial fibrillary acidic protein have led to increased interest into the role of I2BS and I2BS ligands in conditions characterised by marked gliosis. The number of I2BS has been shown to increase in Alzheimer's disease post mortem, and it has also been suggested that I2BS may be a marker for the severity and malignancy of human glioblastomas.

The lack of suitable imaging tools for the I2BS has meant that information regarding the number and distribution of I2BS in the brain has come from preclinical species and in vitro post-mortem studies. The recent development of [11C]BU99008 as a suitable PET ligand to quantify I2BS in vivo, enables the direct quantification of I2BS availability and regional distribution in the living human brain. In this study the investigators plan to utilise [11C]BU99008 to quantify the regional brain availability of I2BS in the human brain in vivo using PET.

DETAILED DESCRIPTION:
This study will consist of three parts; Part A, B and C. Part A will involve up to 10 healthy subjects in order to determine the number and regional location of I2BS in healthy human brain following administration of [11C]BU99008. In Part B up to 6 healthy subjects will be recruited to provide sufficient PET data to quantify the intra- and inter-subject variability in the regional expression of I2BS in healthy human brain. Finally, in Part C up to 6 healthy subjects will be recruited in order to determine the distribution of I2BS in the whole body following administration of [11C]BU99008.

The three parts of this study will be conducted in series, and only if each part is successful will the investigators progress to the next. This will allow us to terminate the study early, and hence prevent the un-necessary exposure of participants to ionising radiation, if the emerging data shows a clear No-go decision to progress with this PET ligand.

Potential participants that pass the initial telephone screen will be invited to a screening visit where their eligibility to take part in the study will be determined and informed consent taken. This will be at the Imperial CRF and Imanova Ltd. The screening will consist of an interview where the study will be discussed and explained. The participants'understanding of the procedure, requirements and commitments confirmed and any questions answered before informed consent taken. In addition to this interview the participants personal details and demographics will be recorded and a psychiatric and medical history taken as well as the following:

* Semi-structured interviews/questionnaires will be completed: Mini International Neuropsychiatric Interview 5 (MINI 5), Cognitive diagnostic test for dementia (CAMCOG)
* A medical examination and blood taken for clinical laboratory testing.
* A structural MRI.
* Review of your medical history and current state of health, including questions about psychiatric symptoms and your use of prescription and non-prescription drugs, as well as your use of illegal drugs and alcohol.
* Physical examination such as measurements of blood pressure and heart rate, ECG.
* Collecting a urine sample to check for presence of drugs.
* Alcohol breath test.
* An "Allen's Test" will be performed to check the blood supply to your hand.
* Other questionnaires: Hospital Anxiety and Depression Scale (HADS), Eysenck personality (revised) (EPQ-R25), Spielberger Trait Anxiety Inventory (STAI), and MRI safety Participants that are eligible will then be invited to take part in the study, either Parts A, B or C as detailed below.

Below is the intended schedule of scanning for this study. However, if for some reason it is necessary to cancel or suspend a scan due to radioligand production failure, scanner failure, etc., the participant will be asked to return on another day to. This will only happen if they have not had the radioligand administered by the time the study is suspended. As detailed below cannulae will be introduced to collect blood for various analysis on the study days (approximately 120 mL). The blood collected for any one participant will not exceed 500 mL for the entire study.

Part A

This will be a study in healthy volunteers, and will involve up to 10 healthy human subjects, with each subject required to receive up to three PET scans over two study days:

* Scanning Day 1; Morning - baseline scan with [11C]BU99008 alone to determine the total number of binding sites (total, PET signal).
* Scanning Day 1; Afternoon - blocking scan with [11C]BU99008 in combination a single dose of idazoxan (I2BS block) • Scanning Day 2; All day - blocking scan with [11C]BU99008 in combination a single dose of isocarboxazid (MAO block) The combination of all three scans will allow us dissect out the regional contribution of the I2BS and MAO components to the [11C]BU99008 specific signal, in order to get an accurate determination of the number of I2BS in different brain regions. The investigators are confident that any component of the [11C]BU99008 signal due to MAO will be negligible. If this is confirmed the second scanning day will be discontinued. This adaptive approach will allow us to minimise unnecessary exposure of the participants to ionising radiation and study medication.

Scanning day 1 - The participants will arrive at Imanova's scanning facility in the Burlington Danes Building, Hammersmith Hospital in the early morning. The exact time will be determined by the logistical constraints for two productions of [11C]BU99008. On arrival, participants will be asked if they agree to carry on participating in the study and their general health and compliance to study specific restrictions assessed by interview, urine drugs of abuse screen and breathalyser. Once it is confirmed they are eligible to proceed, they will be undergo the various procedures for that day.

The participants will be cannulated in the radial artery and have a venous cannula inserted in the forearm or cubital veins. The arterial cannula is required for arterial blood sampling throughout the scan. A venous cannula is required for the administration of [11C]BU99008. If the on-going analysis indicates that arterial blood samples are not required for the analysis of [11C]BU99008, then these samples will not be taken from future subjects participating in this study and the cannula not implanted.

Baseline subjective and objective measures will be taken before they are prepared and positioned in the scanner for PET scan 1. The scan will be approximately 120 min in length, during which time heart rate and blood pressure will be monitored. At the end of the scan, the participants will be removed and another set of subjective and objective measures taken. They will be given an acute dose of idazoxan (up to 80 mg; p.o.) about 120 min before the start of PET scan 2 and another round of subjective and objective measures and arterial blood samples taken as in PET scan 1. At the end of PET scan 2, the participant will be removed from the scanner, any indwelling cannulae removed, a final round of subjective and objective measures recorded, and their fitness to be sent home assessed by the attending physician. When they are fit to leave they will be sent home in a taxi.

Scanning day 2 - The day will be similar to scanning day 1 but there will only be the one scan (PET scan 3). Participants will arrive at Imanova's scanning facility in the Burlington Danes Building, Hammersmith Hospital. Unlike scanning day 1 the time of arrival will be flexible, the exact arrival time will be determined by synthesis of the [11C]BU99008 and the most convenient time for the participant. On arrival, participants will be asked if they agree to carry on participating in the study and their general health and compliance to study specific restriction assessed by interview, urine drugs of abuse screen and breathalyser. Once it is confirmed they are eligible to proceed the participants will be cannulated as before (if required). Baseline subjective and objective measures will be taken and they will be administered an acute dose of isocarboxazid (up to 50 mg; p.o.) about 240 min before the start of PET scan 3. A round of subjective and objective measures will be recorded before they are prepared and positioned in the scanner for PET scan 3 (as above). At the end of the scan the participant will be removed from scanner, any indwelling cannulae removed, a final round of subjective and objective measures recorded, and their fitness to be sent home assessed by the attending physician. When they are fit to leave they will be sent home in a taxi.

Part B

This part of the study is to understand how the intra- and inter-subject variability in the I2BS regional density differs in a healthy population. To assess this, up to 6 healthy volunteers will receive two scans of [11C]BU99008 alone, on two separate study days:

* Scanning Day 1 - scan with [11C]BU99008 alone
* Scanning Day 2 - scan with [11C]BU99008 alone The combination of these two scans will enable us to determine both the intra- and inter-subject variability for the expression of the I2BS in a normal population.

On arrival, participants will be asked if they agree to carry on participating in the study. In addition, the general health and compliance of participants to study specific restriction will be assessed by interview, urine drugs of abuse screen and breathalyser. The participants will be cannulated as described above (if required). Baseline subjective and objective measures will be taken prior to preparation and positioning in the scanner for the PET scan. The scan will be approximately 120 min in length during which heart rate and blood pressure will be monitored. In addition, as in Part A, arterial and/or venous blood samples will be taken throughout the scan. At the end of the scan the participants will be removed from the scanner, any indwelling cannulae removed and a final round of subjective and objective measures recorded. At this point the fitness of participants to be sent home will be assessed by the attending physician. When they are fit to leave they will be sent home in a taxi.

Part C This part of the study is to determine the whole body bio-distribution of the I2BS in healthy humans. Up to 6 healthy subjects will be enrolled into this part of the study to determine the number and distribution of the I2BS in a variety of tissues and organs. Each participant will receive one whole body PET scan of [11C]BU99008. This whole body scan will enable us to determine how the I2BS is distributed in tissues and organs in addition to the brain. Participants in this part of the study will receive only one PET scan on their single study visit. On arrival participants will be asked if they agree to carry on participating in the study. In addition, the general health and compliance of participants to study specific restriction will be assessed by interview, urine drugs of abuse screen and breathalyser. The participants will be cannulated as above. Baseline subjective and objective measures will be taken prior to preparation and positioning in the scanner for the PET scan. The scan will be probably be 240 min in length (two, 2hr sessions with a break in-between) during which heart rate and blood pressure will be monitored. In addition, as in Parts A and B, arterial blood samples will be taken throughout the scan. Unlike the PET scans for Parts A & B this scan will occur over the whole body scan and not just the brain. At the end of the scan the participants will be removed from the scanner, any indwelling cannulae removed and a final round of subjective and objective measures recorded. At this point their fitness to be sent home will be assessed by the attending physician. When they are fit to leave they will be sent home in a taxi.

ELIGIBILITY:
Inclusion Criteria:

* Male between 40 and 65 years at the time of signing the informed consent Non-smoker
* Willing to comply with protocol and lifestyle restrictions
* Excellent understanding of English (for questionnaires)
* Subject is ambulant and capable of attending a PET scan visit as an outpatient.
* Subjects with female partners of child-bearing potential must agree to use one of the contraception methods permitted by the study. This criterion must be followed from after the first PET Scan until after the follow-up contact.
* Adequate collateral flow to the radial and ulnar arteries in both hands as determined by an Allen's test.
* Body weight ≥50 kg.
* Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, objective physiological measures, previous laboratory studies, and other tests.
* Successful completion of the CAMCOG.

Exclusion Criteria:

* Current or past history of major psychiatric disorder
* Current or past history of substance use disorder
* Clinically significant brain injury or abnormality
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of or suffers from claustrophobia or subject feels unable to lie flat and still on their back for a period of up to 2 hours in the PET/CT scanner.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations or occupational exposure resulting in radiation exposure greater than 10 mSv over the past 3 years or greater than 10 mSv in a single year including the proposed study. Clinical exposure from which the subject receives a direct benefit is not included in these calculations.
* Previous inclusion in a research and/or medical protocol involving study medication within the last 3 months
* In the opinion of the study team they are unlikely to comply with the study protocol and restrictions that it imposes.
* Contraindications for subjects undergoing an MR scan (including but not limited to metal implants pacemakers, etc.)

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Nutt, MD, Principal Investigator — Director of Centre for Neuropsychopharmacology, Imperial College London
Locations (1):
- Centre for Neuropsychopharmacology; Division of Brain Sciences; Imperial College London; Burlington Danes Building; Hammersmith Hospital campus; 160 Du Cane Road, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Regional Density and Distribution of I2BS in Healthy Human Brain (1TCM Model)
Description: The determination of the regional density and distribution of the I2BS in human brain of healthy volunteers. The output parameter used to determine this will be derived from the most appropriate PET pharmacokinetic model for this ligand in human e.g. Total Volume of Distribution (VT) or Binding Potential (BP).
  Regional time-activity data were generated from arterial plasma input functions corrected for metabolites using the most appropriate model to derive the outcome measure VT (regional distribution volume). All image processing and kinetic analyses were performed in MIAKAT. The Akaike model selection criteria were used to determine the most appropriate model to describe these data.
  The calculated criteria for the three main models are: one-tissue (1TCM) and two-tissue (2TCM) compartmental models, and multilinear analysis model (MA).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 18
mL/cm^3
  Whole Brain | 44.5 (6.1)
  Cerebellum | 39.3 (6.2)
  Brain stem | 62.7 (9.1)
  Occipital lobe | 38.6 (6.5)
  Insula | 63.3 (9.0)
  Frontal lobe | 41.6 (5.9)
  Cingulate | 58.3 (8.6)
  Parietal lobe | 39.2 (5.8)
  Amygdala | 89.8 (15.2)
  Hippocampus | 68.4 (11.4)
  Striatum | 102.7 (17.8)
  Thalamus | 75.3 (11.0)

2. Secondary Outcome: Intra- and Inter-Subject Variability in Brain Expression of Imidazoline 2 Binding Sites, Measured Using Coefficient of Variability (%COV), Determined From Either Total Volume of Distribution (VT) or Binding Potential (BP).
Description: To evaluate the variability in the regional brain expression of I2BS within and between subjects using coefficient of variability (%COV). The %COV will be obtained from the most appropriate I2BS expression measures either Total Volume of Distribution (VT) or Binding Potential (BP).
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Peripheral Distribution of Imidazoline 2 Binding Sites Using Either Total Volume of Distribution (VT) or Binding Potential (BP)
Description: To evaluate the distribution of I2BS in the human body. The output parameter used to determine this will be derived from the most appropriate PET pharmacokinetic model for this ligand in human e.g. Total Volume of Distribution (VT) or Binding Potential (BP).
Time Frame: 1 year
Reporting Status: Not Posted

4. Primary Outcome: Determination of the Regional Density and Distribution of I2BS in Healthy Human Brain (2TCM Model)
Description: as for outcome 1
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 18
mL/cm^3
  Whole Brain | 48.8 (7.9)
  Cerebellum | 41.9 (6.9)
  Brain stem | 66.4 (10.1)
  Occipital lobe | 42.7 (8.6)
  Insula | 67.7 (11.8)
  Frontal lobe | 45.7 (7.9)
  Cingulate | 62.2 (9.7)
  Parietal lobe | 43.6 (8.7)
  Amygdala | 94.6 (20.3)
  Hippocampus | 77.7 (24.2)
  Striatum | 105.7 (21.0)
  Thalamus | 80.0 (14.1)

5. Primary Outcome: Determination of the Regional Density and Distribution of I2BS in Healthy Human Brain (MA Model)
Description: as for outcome 1
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 18
mL/cm^3
  Whole Brain | 44.8 (6.1)
  Cerebellum | 39.6 (6.2)
  Brain stem | 63.2 (9.2)
  Occipital lobe | 38.8 (6.5)
  Insula | 63.9 (9.1)
  Frontal lobe | 42.0 (5.9)
  Cingulate | 58.8 (8.6)
  Parietal lobe | 39.5 (5.9)
  Amygdala | 91.1 (15.1)
  Hippocampus | 69.1 (11.5)
  Striatum | 104.2 (17.6)
  Thalamus | 76.0 (11.1)

ADVERSE EVENTS:
Arm/Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes